CLINICAL TRIAL: NCT04637828
Title: Cure COVID: A Prospective, Controlled, Randomized Study to Compare the Efficacy of GNS561 Versus Standard of Care in Patients With SARS-CoV-2 (COVID-19) Infection
Brief Title: A Study to Compare the Efficacy of GNS561 Versus Standard of Care in Patients With SARS-CoV-2 (COVID-19) Infection
Acronym: CureCovid-2019
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genoscience Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GNS561-CL-I-Q-0291
Record Dates: First submitted 2020-11-17; First posted 2020-11-20 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2020-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: open-label, controlled, randomized phase 2 study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GNS561 plus standard of care (Experimental): All patients in this Arm will be treated with 200mg oral capsule of GNS561, once a day, for 10 days and with any necessary measures based on the patient's condition and at the investigator's discretion and routine practices.
  Interventions: Drug: GNS561
- standard of care (No Intervention): All patients in this Arm will be treated with any necessary measures based on the patient's condition and at the investigator's discretion and routine practices.

INTERVENTIONS:
Drug: GNS561 — study drug
  Arms: GNS561 plus standard of care

SUMMARY:
This is a multicenter, open-label, controlled, randomized phase 2 study designed to evaluate the safety and efficacy profile of GNS561 in patients with COVID-19.

DETAILED DESCRIPTION:
Patients will be treated either with oral GNS561 plus standard of care or only standard of care. All patients in experimental arm will be treated for ten days. Study drug will be provided as oral capsules containing 200 mg of GNS561. Patients will be followed-up during hospitalization and after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of COVID-19 (diagnostic test performed in a certified laboratory).
* Clinical status: Hospitalized for moderate COVID-19 with News2 score between 5 and 6

Exclusion Criteria:

* Patient known to have intolerance or hypersensitivity to chloroquine or any quinoline derivates (quinine, tafenoquine, hydroxychloroquine, mefloquine).
* History of QT prolongation (QTc ≥ 500 ms) or QTc ≥ 500msec at screening or bradycardia < 50/mn
* Current use of loop diuretics and potassium supplementation or documented history of hypokalemia or hypokalemia < 3.5mmol/l at screening
* Prior allogeneic bone marrow transplantation or solid organ transplant in the past.
* Pregnant or breastfeeding patient, or expecting to conceive children within the projected duration of the trial, starting with the screening visit through 6 months after the last dose of study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — age 18 or older at the time of enrolment for women and age 60 or older at the time of enrolment for men.
Enrollment: 178 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
number and proportion of participants, per randomized group, with a loss of one or two grades of National Early Warning Score (NEWS2) score at day-7 compared to baseline | 7 days
  severe stage at baseline to medium or low stage at day-7 or medium stage at baseline to low stage at day-7

SECONDARY OUTCOMES:
the 28-day survival rate | 28 days
  the crude proportion of patients still alive 28 days after randomization
the rate of intensive care unit admission | 14 days
  to 14 days from randomization
the rate of nasopharyngeal swab negativation at D7, D14 and D28 | 7 days, 14 days and 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Genoscience Pharma, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided